CLINICAL TRIAL: NCT06306131
Title: A Phase II Study to Evaluate the Delay in Ovulation Following Oral Levonorgestrel Plus Meloxicam Compared to Placebo in Obese But Normal Menstruating Women
Brief Title: Phase II Study of Ovulation in Obese Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InnovaGyn, Inc. (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IG-23-002; 1R43HD107861-01A1 (NIH)
Record Dates: First submitted 2023-12-18; First posted 2024-03-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Prevention
Keywords: Female; Hormonal contraception; Emergency Contraception; levonorgestrel; meloxicam
MeSH Terms: interventions — Levonorgestrel; Meloxicam

STUDY DESIGN:
Intervention Model Description: Placebo controlled in first cycle with levonorgestrel plus meloxicam in second menstrual cycle.
Who Masked: Outcomes Assessor
Masking Description: The intervention will be masked to the laboratory preforming the analysis of the urinary metabolites. The statistician, clinicians, coordinators and participants will be aware of the medication being studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo is calcium carbonate 750 milligram (mg) known as TUMS. Each participant will take one tablet orally and repeat 48 hours later.
  Interventions: Other: calcium carbonate 750 milligram
- Levonorgestrel plus meloxicam (Active Comparator): The active comparator is levonorgestrel 1.5 milligram (mg) and meloxicam 15 milligram (mg) taken together orally and repeated 48 hours later.
  Interventions: Drug: Levonorgestrel 0.15 milligram; Drug: Meloxicam 15 milligram

INTERVENTIONS:
Drug: Levonorgestrel 0.15 milligram — The study design is an open label randomized single blind clinical trial in which each participant will receive placebo two tablets 48 hours apart in their first menstrual cycle and then levonorgestrel plus meloxicam 48 hours apart in their subsequent menstrual cycle. We will compare the interval from taking the first dose of medication to the development of a functioning corpus luteum based on the shift in the ratio of urinary estrone-3-glucuronide(EC) / pregnanediol-3-glucuronide (PDG).
  Other Names: Plan B one Step
  Arms: Levonorgestrel plus meloxicam
Drug: Meloxicam 15 milligram — The study design is an open label randomized single blind clinical trial in which each participant will receive placebo two tablets 48 hours apart in their first menstrual cycle and then levonorgestrel plus meloxicam 48 hours apart in their subsequent menstrual cycle. We will compare the interval from taking the first dose of medication to the development of a functioning corpus luteum based on the shift in the ratio of urinary estrone-3-glucuronide(EC) / pregnanediol-3-glucuronide (PDG).
  Other Names: Mobic
  Arms: Levonorgestrel plus meloxicam
Other: calcium carbonate 750 milligram — The study design is an open label randomized single blind clinical trial in which each participant will receive placebo two tablets 48 hours apart in their first menstrual cycle and then levonorgestrel plus meloxicam 48 hours apart in their subsequent menstrual cycle. We will compare the interval from taking the first dose of medication to the development of a functioning corpus luteum based on the shift in the ratio of urinary estrone-3-glucuronide(EC) / pregnanediol-3-glucuronide (PDG).
  Other Names: TUMS
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare the delay in ovulation between placebo to levonorgestrel plus meloxicam in obese women with normal menses. The main questions it aims to answer are:

1. Ovulation will be delayed by ≥7 days following the first dose of levonorgestrel plus meloxicam compared to ovulation within 3 days following the first dose of placebo.
2. There will be no difference in unscheduled vaginal bleeding or adverse events between the two treatments [placebo versus levonorgestrel plus meloxicam].

Participants will:

* undergo two treatment cycles the 1st uses placebo and the 2nd is levonorgestrel plus meloxicam,
* maintain daily diary logs for adverse events, unscheduled bleeding, and onset, cessation, and amount of menstrual bleeding,
* collect daily first morning voided urine from menstrual day 9 to 24,
* undergo transvaginal ultrasound for ovarian follicle development on menstrual days 9, 11,13 and 14.
* allow a blood sample to be drawn on days with ultrasound scans.
* Take 1st placebo and levonorgestrel plus meloxicam under observation when dominant ovarian follicle is 17 ±1.0 millimeters (mm) in diameter and 2nd dose 48 hours later.

Researchers will compare the placebo cycle to levonorgestrel plus meloxicam to see if ovulation is delayed, there is unscheduled vaginal bleeding, menstrual onset is delayed or there is an abnormal amount or duration of menses, there is any difference in treatment emergent side effects and any change in vital signs

DETAILED DESCRIPTION:
We will perform a single site clinical trial in obese women not at risk of pregnancy aged 18 to 40. We will screen to enroll and complete 22 participants. Each participant after signing an Informed Consent and meeting all inclusion and exclusion criteria will be enrolled on menstrual day 9-10 of a subsequent menstrual cycle following a negative urine pregnancy test. Each participant will be asked to collect a first morning voided urine sample beginning on menstrual day 9 and completing 15 days later on menstrual day 24. The participant will undergo a transvaginal ultrasound on menstrual days 9-10, 12, 13 and day 14 to determine ovarian follicle diameters in two planes frontal and sagittal using transvaginal ultrasound. When the largest follicle diameter is 17±1.0 millimeters (mm) the participant will be given the intervention: placebo in the 1st cycle and levonorgestrel plus meloxicam in the 2nd cycle followed by a second dose of each intervention 48 hours later. The ovarian follicle dimension of 17 mm occurs in the middle of the woman's window of fertility which is the four days preceding plus the day of ovulation. We anticipate that ovulation will take place within 3 days after the first placebo dose in 90% of the participants and will be delayed ≥7 days following the first dose of levonorgestrel plus meloxicam in ≥80% of the participants. The primary outcome is the delay in days from the first dose to evidence of ovarian corpus luteum formation which follows ovulation. All urine samples from the same participant will be analyzed in one assay for estrogen and progesterone metabolites to reduce inter-assay variability. The primary outcome will be delay of ovulation based on changes in the ratio of the urinary metabolites in obese women between placebo and active treatment. Secondary outcomes (exploratory) are a) safety parameters vital signs consisting of blood pressure and pulse obtained at each visit, b) adverse events, unscheduled bleeding, and changes in menstrual bleeding captured by the participant using a daily diary card. She will be instructed to write down any symptoms or problem along with medication taken both study drug and any other medication. Any treatment adverse event considered to be serious will be reported to the local institutional review board and the Food and Drug Administrating within 72 hours of our being made aware of the problem. The occurrence, percentage, and relationship to study drug of minor and moderate adverse events will be noted and categorized using Medical Dictionary for Regulatory Activates (MedRA) adverse event classification and listed in all reports and publications.

Each participant will be involved for a study period of approximately 2.5 months or 75 days. Each participant will undergo a complete history and physical evaluation at entry and a brief interim history and physical evaluation at exit with height and weight at entry. Mean and standard deviation of all vital signs before and after treatment, menstrual bleeding changes and treatment emergent adverse events will be compiled and listed in all reports and publications.

ELIGIBILITY:
Inclusion Criteria:

1. Female in good general health with no chronic medical conditions that result in periodic exacerbations that require significant medical care.
2. Age between 18 to 40 years inclusive at time of enrollment.
3. BMI ≥30 kg/m² and no recent rapid weight loss or gain.
4. Intact uterus with both ovaries intact.
5. Papanicolaou test within American Society for Colposcopy and Cervical Pathology (ASCCP), or American College of Obstetricians and Gynecologists (ACOG) guidelines such that additional testing or evaluation will not be required during the study period. If there is no copy of a recent Papanicolaou test and the subject is 21 years or older a Papanicolaou test should be done during the screening visit.
6. Regular menstrual cycles with an interval of 24 to 32 days:

   1. If postpartum or post-second trimester abortion, she must have 2 spontaneous menses prior to enrollment.
   2. If the subject has had a first trimester pregnancy loss or abortion, she must have one spontaneous menses prior to enrollment.
7. Have a negative urine pregnancy test on menstrual cycle day 9 pre-treatment visit.
8. Not at risk of pregnancy for the duration of the study defined as heterosexually abstinent, prior female or male permanent contraception, non-hormonal intrauterine device or willing to use a non-hormonal barrier contraceptive method with each act of intercourse until study exit.
9. Subject is willing and able in the Investigators opinion of complying with protocol requirements.
10. Subject is willing to collect daily first morning urines and store them until brought to the study site.
11. Lives within the study catchment area or a reasonable distance from the study site.
12. Understands and signs the IRB approved informed consent prior to undergoing any screening assessment.
13. Agrees not to participate in any other clinical trials during the course of this study.
14. Screening serum progesterone level greater than 3 ng/ml.-

Exclusion Criteria:

1. Known hypersensitivity or contraindications to progestins.
2. Abnormal transvaginal ultrasound or safety laboratory results evaluated during the screening period recognized as clinically significant by the investigator or medically qualified designee.
3. Known or suspected alcohol or marijuana abuse.
4. Undiagnosed abnormal genital bleeding.
5. Undiagnosed vaginal discharge, lesions or abnormalities.
6. Women with a history of genital herpes can be included if the outbreaks are infrequent. Antiviral prophylaxis is allowed.
7. Uncontrolled Thyroid disorder.
8. Current use of hormonal contraception or a levonorgestrel releasing intrauterine device.
9. Use of a long-acting injectable hormonal contraceptive within the past 6 months unless has had at least one spontaneous menstrual cycle (two menstrual bleeding episodes) since the last injection.
10. Breastfeeding women or those who have not had a spontaneous menstrual bleed since discontinuing breastfeeding.
11. Women who plan a major surgical procedure during the study.
12. Women who plan to become pregnant during their participation in the study.
13. Women who smoke >15 cigarettes per day or who use >1 mL/day of nicotine-containing liquid for electronic cigarettes.
14. Current or history of ischemic heart disease or stroke while pregnant or during use of hormonal contraception.
15. Current or past deep vein thrombosis or thromboembolic disorder.
16. Personal or family history of thrombophilia
17. History of retinal vascular lesions or partial or complete loss of vision.
18. Known or suspected carcinoma of the breast, endometrium, or other suspected progestin sensitive neoplasia.
19. History of other carcinomas excluding basal cell cancers unless in remission for > 5 years.
20. Current or past medically diagnosed severe depression unless the potential participant is on stable medication or in the opinion of the Principal Investigator could be exacerbated using a hormonal contraceptive.
21. History of headaches with focal neurologic symptoms.
22. Have a current need for exogenous hormones or therapeutic anticoagulants.
23. History of cholestatic jaundice of pregnancy or jaundice with prior steroid hormone use.
24. Other benign or malignant liver tumors or active liver disease.
25. Systolic BP ≥145 mm Hg and/or diastolic BP ≥96 mm Hg after 5 -10 minutes of rest in a sitting position. If the initial BP values are above these cut-offs, a total of 3 measurements may be taken and the results averaged. If the averaged BP is below the cut-off levels, the participant may be allowed into the study. Hypertension that is treated and controlled may be allowed based on the Investigator's discretion.
26. Clinically significant abnormal serum chemistry value based on the Investigator's judgement.
27. Participation in another clinical trial involving an investigational drug or device within the past two months before anticipated enrollment or is planning to participate in another clinical study during this study.
28. Use of any liver enzyme inducers or plans to use such medication during the study.
29. Known HIV infection.
30. History of a gastrointestinal ulcer or bleeding.
31. Women who are using medication on the Exclusionary medication list (See Appendix).
32. Have issues or concerns, in the opinion of the Investigator, that may compromise the study or confound the reliability of compliance and information that is required in this study.
33. Have a known hypersensitivity to either levonorgestrel or a non-steroidal anti-inflammatory drug.
34. Use of any medication that could interfere with the metabolism of a hormonal contraceptive or the non-steroidal anti-inflammatory drugs or any drug that falls in FDA Pregnancy and Lactation narrative subsections (Formerly Category D or X medications).
35. Be a site member with delegated study responsibilities or a family member of, or have a close relationship with, a site staff member who will be delegated study responsibilities.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Designated as female at birth.
Enrollment: 22 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Interval from first dose to evidence of ovulation. | The interval is estimated to be 3 days from first dose to evidence of ovulation with placebo and 7 days following active treatment.
  An ovarian follicle diameter of 17 mm is used to take the first dose of medication. Daily morning urine samples are analyzed for estrone-3-glucronide and pregnanediol-3-glucuronide. Changes in the ratio of these two metabolites is indicative of ovulation termed the follicular luteal shift. The interval from first dose to follicular luteal shift is estimated to be 3 days. The active treatment will be given when the ovarian follicle diameter is also 17 mm. The outcome is estimated to be a delay of 7+ days from 1st dose to the follicular luteal shift or ovulation

SECONDARY OUTCOMES:
Change in blood pressure | The blood pressure is monitored at screening and from menstrual day 9 to 24 in each of two treatment cycles.
  Sitting blood pressure in millimeters mercury (mm Hg) will be recorded at each visit. The outcome is a significant change in systolic, and diastolic blood pressure in millimeters of mercury during each treatment.
Change in Pulse | Pulse rate is measured at all visits throughout the study
  Pulse measured in beats per minute at the wrist

OTHER OUTCOMES:
Unscheduled endometrial bleeding and changes in interval, amount and duration of menstrual bleeding. | Daily diary cards will be kept by each participant beginning menstrual day 9 of first cycle. Diary cards will be returned at the exit visit within two weeks of the final (second) menstrual period.
  Each participant will enter on daily diary cards any unscheduled vaginal bleeding, onset and duration of menstrual period and amount of menstrual blood loss. These changes if any will be compared between placebo and levonorgestrel plus meloxicam.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lukes, MD, Principal Investigator — Carolina Woman's Research and Wellness Center
Locations (1):
- Carolina Women's Research and Wellness Center, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Raymond EG, Shochet T, Drake JK, Westley E. What some women want? On-demand oral contraception. Contraception. 2014 Aug;90(2):105-10. doi: 10.1016/j.contraception.2014.04.008. Epub 2014 Apr 21. PMID 24835831
- [Result] Daniels K, Mosher WD. Contraceptive methods women have ever used: United States, 1982-2010. Natl Health Stat Report. 2013 Feb 14;(62):1-15. PMID 24988816
- [Result] Moreau C, Cleland K, Trussell J. Contraceptive discontinuation attributed to method dissatisfaction in the United States. Contraception. 2007 Oct;76(4):267-72. doi: 10.1016/j.contraception.2007.06.008. Epub 2007 Aug 28. PMID 17900435
- [Result] Trussell J. Contraceptive failure in the United States. Contraception. 2004 Aug;70(2):89-96. doi: 10.1016/j.contraception.2004.03.009. PMID 15288211
- [Result] Simmons RG, Sanders JN, Geist C, Gawron L, Myers K, Turok DK. Predictors of contraceptive switching and discontinuation within the first 6 months of use among Highly Effective Reversible Contraceptive Initiative Salt Lake study participants. Am J Obstet Gynecol. 2019 Apr;220(4):376.e1-376.e12. doi: 10.1016/j.ajog.2018.12.022. Epub 2018 Dec 18. PMID 30576664
- [Result] Venners SA, Liu X, Perry MJ, Korrick SA, Li Z, Yang F, Yang J, Lasley BL, Xu X, Wang X. Urinary estrogen and progesterone metabolite concentrations in menstrual cycles of fertile women with non-conception, early pregnancy loss or clinical pregnancy. Hum Reprod. 2006 Sep;21(9):2272-80. doi: 10.1093/humrep/del187. Epub 2006 Jun 23. PMID 16798842
- [Result] Bradley SEK, Polis CB, Bankole A, Croft T. Global Contraceptive Failure Rates: Who Is Most at Risk? Stud Fam Plann. 2019 Mar;50(1):3-24. doi: 10.1111/sifp.12085. Epub 2019 Feb 21. PMID 30791104
- [Result] Pace LE, Dusetzina SB, Keating NL. Early Impact Of The Affordable Care Act On Oral Contraceptive Cost Sharing, Discontinuation, And Nonadherence. Health Aff (Millwood). 2016 Sep 1;35(9):1616-24. doi: 10.1377/hlthaff.2015.1624. PMID 27605641
- [Result] Duffy DM, Ko C, Jo M, Brannstrom M, Curry TE. Ovulation: Parallels With Inflammatory Processes. Endocr Rev. 2019 Apr 1;40(2):369-416. doi: 10.1210/er.2018-00075. PMID 30496379
- [Result] Croxatto HB, Brache V, Pavez M, Cochon L, Forcelledo ML, Alvarez F, Massai R, Faundes A, Salvatierra AM. Pituitary-ovarian function following the standard levonorgestrel emergency contraceptive dose or a single 0.75-mg dose given on the days preceding ovulation. Contraception. 2004 Dec;70(6):442-50. doi: 10.1016/j.contraception.2004.05.007. PMID 15541405
- [Result] Devoto L, Fuentes A, Palomino A, Espinoza A, Kohen P, Ranta S, von Hertzen H. Pharmacokinetics and endometrial tissue levels of levonorgestrel after administration of a single 1.5-mg dose by the oral and vaginal route. Fertil Steril. 2005 Jul;84(1):46-51. doi: 10.1016/j.fertnstert.2005.01.106. PMID 16009156
- [Result] Brache V, Cochon L, Deniaud M, Croxatto HB. Ulipristal acetate prevents ovulation more effectively than levonorgestrel: analysis of pooled data from three randomized trials of emergency contraception regimens. Contraception. 2013 Nov;88(5):611-8. doi: 10.1016/j.contraception.2013.05.010. Epub 2013 May 22. PMID 23809278
- [Result] Duffy DM. Novel contraceptive targets to inhibit ovulation: the prostaglandin E2 pathway. Hum Reprod Update. 2015 Sep-Oct;21(5):652-70. doi: 10.1093/humupd/dmv026. Epub 2015 May 29. PMID 26025453
- [Result] Glasier A, Cameron ST, Blithe D, Scherrer B, Mathe H, Levy D, Gainer E, Ulmann A. Can we identify women at risk of pregnancy despite using emergency contraception? Data from randomized trials of ulipristal acetate and levonorgestrel. Contraception. 2011 Oct;84(4):363-7. doi: 10.1016/j.contraception.2011.02.009. Epub 2011 Apr 2. PMID 21920190
- [Result] Glasier A. Emergency contraception: clinical outcomes. Contraception. 2013 Mar;87(3):309-13. doi: 10.1016/j.contraception.2012.08.027. Epub 2012 Oct 4. PMID 23040128
- [Result] Gemzell-Danielsson K, Berger C, P G L L. Emergency contraception -- mechanisms of action. Contraception. 2013 Mar;87(3):300-8. doi: 10.1016/j.contraception.2012.08.021. Epub 2012 Oct 29. PMID 23114735
- [Result] Festin MP, Bahamondes L, Nguyen TM, Habib N, Thamkhantho M, Singh K, Gosavi A, Bartfai G, Bito T, Bahamondes MV, Kapp N. A prospective, open-label, single arm, multicentre study to evaluate efficacy, safety and acceptability of pericoital oral contraception using levonorgestrel 1.5 mg. Hum Reprod. 2016 Mar;31(3):530-40. doi: 10.1093/humrep/dev341. Epub 2016 Jan 31. PMID 26830816
- [Result] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Result] Jesam C, Salvatierra AM, Schwartz JL, Croxatto HB. Suppression of follicular rupture with meloxicam, a cyclooxygenase-2 inhibitor: potential for emergency contraception. Hum Reprod. 2010 Feb;25(2):368-73. doi: 10.1093/humrep/dep392. Epub 2009 Nov 19. PMID 19933235
- [Result] Bata MS, Al-Ramahi M, Salhab AS, Gharaibeh MN, Schwartz J. Delay of ovulation by meloxicam in healthy cycling volunteers: A placebo-controlled, double-blind, crossover study. J Clin Pharmacol. 2006 Aug;46(8):925-32. doi: 10.1177/0091270006289483. PMID 16855077
- [Result] Massai MR, Forcelledo ML, Brache V, Tejada AS, Salvatierra AM, Reyes MV, Alvarez F, Faundes A, Croxatto HB. Does meloxicam increase the incidence of anovulation induced by single administration of levonorgestrel in emergency contraception? A pilot study. Hum Reprod. 2007 Feb;22(2):434-9. doi: 10.1093/humrep/del369. Epub 2006 Sep 15. PMID 16980507
- [Result] Santoro N, Crawford SL, Allsworth JE, Gold EB, Greendale GA, Korenman S, Lasley BL, McConnell D, McGaffigan P, Midgely R, Schocken M, Sowers M, Weiss G. Assessing menstrual cycles with urinary hormone assays. Am J Physiol Endocrinol Metab. 2003 Mar;284(3):E521-30. doi: 10.1152/ajpendo.00381.2002. Epub 2002 Nov 19. PMID 12441312
- [Result] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

DOCUMENTS (1):
  • Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT06306131/ICF_000.pdf